CLINICAL TRIAL: NCT06078761
Title: A Prospective Study of the Healthy Eating and Active Lifestyle (HEAL): Breast Cancer Program on Survivorship Outcomes
Brief Title: Healthy Eating and Active Lifestyle (HEAL): Breast Cancer Program Outcomes
Acronym: HEAL BC
Status: Recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 2056943
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Healthy Eating Active Lifestyle (HEAL) Program — Evidence-based lifestyle medicine program for cancer survivors

SUMMARY:
The goal of this single-group prospective study is to examine the impact of the Healthy Eating and Active Lifestyle (HEAL) Breast Cancer program on participants' perceived stress, biometrics, basic labs, lifestyle behaviors, self-efficacy, mental health, and quality of life.

Participants will participate in an 8-week program of 90-minute virtual sessions each week to decrease risk of cancer recurrence. Program participants can choose to participate in the research study which will include data collection (surveys, biometrics, basic labs). The data collection will occur at four timepoints - baseline prior to program start, post-program, 3 month follow-up, and 6 month follow-up.

DETAILED DESCRIPTION:
The study will include 45 subjects recruited from AdventHealth Medical Group in the HEAL Breast Cancer Program that consent to participate in the research study. The research study will include data collection along with the program participation. Patients who decline participation in the research study are able to participate in the HEAL Breast Cancer Program. The program sessions will be conducted virtually via Zoom by Dr. Amber Orman, a breast cancer physician board certified in radiation oncology and lifestyle medicine. There are eight program sessions, one per week, each lasting 90-minutes. The survey package includes nine questionnaires and is expected to take 60 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old
2. Diagnosis of breast cancer
3. Enrolled in the HEAL: Breast Cancer Program
4. Able to speak, read, and understand English fluently
5. Willing and able to provide informed consent
6. Willing and able to comply with all study procedures and requirements for the duration of the study

Exclusion Criteria:

1. Not willing or able to provide informed consent
2. Not willing or able to comply with all study procedures and requirements for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors recruited from the AdventHealth Medical Group that were referred to attend the Healthy Eating and Active Lifestyle Breast Cancer Program.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline, Week 8, 3-month follow up, 6-month follow up
  PSS-10 is a ten item questionnaire covering the last month using 5 point Likert scale with 0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Fairly often, 4 = Very often.

SECONDARY OUTCOMES:
mini-Eating Assessment Tool (mini-EAT) | Baseline, Week 8, 3-month follow up, 6-month follow up
  mini-EAT is a 9-item validated brief dietary screener where participants indicate how often they eat food groups with 9 response options: I do not eat it at all, Less than 1 serving per week, 1-2 servings per week, 3-4 servings per week, 5-6 servings per week, 1 serving per day, 2-3 servings per day, 4-5 servings per day, 6 or more servings per day
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Baseline, Week 8, 3-month follow up, 6-month follow up
  Godin-Shephard Leisure-Time Physical Activity Questionnaire includes 3 categories that participants indicate number of times in a week they participate
General Self-Efficacy Scale | Baseline, Week 8, 3-month follow up, 6-month follow up
  The GSE includes 10 items with response categories: 1 = not at all true, 2 = hardly true, 3 = moderately true and 4 = exactly true
Generalized Anxiety Disorder - 2 item scale | Baseline, Week 8, 3-month follow up, 6-month follow up
  The GAD-2 is a 2-item scale about the last 2 weeks with response categories: 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day
Patient Health Questionnaire - 2 item | Baseline, Week 8, 3-month follow up, 6-month follow up
  The PHQ-2 is a 2-item scale about the last 2 weeks with response categories: 0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day
Functional Assessment of Cancer Therapy - General - 7-item version | Baseline, Week 8, 3-month follow up, 6-month follow up
  The FACT-G7 is a 7 item scale about the last 7 days with response categories: 0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much
Weight | Baseline, Week 8, 3-month follow up, 6-month follow up
  Weight in kilograms
Body Mass Index | Baseline, Week 8, 3-month follow up, 6-month follow up
  Body Mass Index (BMI)
Blood pressure | Baseline, Week 8, 3-month follow up, 6-month follow up
  Blood pressure both systolic and diastolic
Lipid panel | Baseline, Week 8, 3-month follow up, 6-month follow up
  Standard of care Lipid panel
Comprehensive metabolic panel | Baseline, Week 8, 3-month follow up, 6-month follow up
  Standard of care Comprehensive metabolic panel
Hemoglobin A1C | Baseline, Week 8, 3-month follow up, 6-month follow up
  Standard of care Hemoglobin A1C

CONTACTS AND LOCATIONS:
Overall Officials: Amanda T. Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] 2. Godin, G. (2011). The Godin-Shephard Leisure-Time Physical Activity Questionnaire. The Health & Fitness Journal of Canada, 4(1), 18-22. https://doi.org/10.14288/hfjc.v4i1.82
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Lara-Breitinger KM, Medina Inojosa JR, Li Z, Kunzova S, Lerman A, Kopecky SL, Lopez-Jimenez F. Validation of a Brief Dietary Questionnaire for Use in Clinical Practice: Mini-EAT (Eating Assessment Tool). J Am Heart Assoc. 2023 Jan 3;12(1):e025064. doi: 10.1161/JAHA.121.025064. Epub 2022 Dec 30. PMID 36583423
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Orman A, Johnson DL, Comander A, Brockton N. Breast Cancer: A Lifestyle Medicine Approach. Am J Lifestyle Med. 2020 Apr 26;14(5):483-494. doi: 10.1177/1559827620913263. eCollection 2020 Sep-Oct. PMID 32922233
- [Background] Patel Saxena S. Leveraging Time With Lifestyle-Based Group Visits. Am J Lifestyle Med. 2016 Jun 23;10(5):330-337. doi: 10.1177/1559827616638018. eCollection 2016 Sep-Oct. PMID 30202290
- [Background] 9. Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy Scale. J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs, 35, 37.
- [Background] Yanez B, Pearman T, Lis CG, Beaumont JL, Cella D. The FACT-G7: a rapid version of the functional assessment of cancer therapy-general (FACT-G) for monitoring symptoms and concerns in oncology practice and research. Ann Oncol. 2013 Apr;24(4):1073-8. doi: 10.1093/annonc/mds539. Epub 2012 Nov 7. PMID 23136235